CLINICAL TRIAL: NCT00455039
Title: INST 0514C- A Neoadjuvant Phase II Trial of GW572016 in HER2 Overexpressing Breast Cancer Patients: Biologic Correlative Study
Brief Title: INST 0514C- Biologic Correlative Study: Trial of GW572016 in HER2 Overexpressing Breast Cancer Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This is a duplicate record and the sponsor has submitted under NCT00206427.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0514C
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: neoadjuvant; HER2; Breast; lapatinib; GSK
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GW572016 1500mg (Experimental): patients received GW572016 1500mg daily
  Interventions: Drug: GW572016

INTERVENTIONS:
Drug: GW572016 — Dose: 1500 mg daily

SUMMARY:
Neoadjuvant chemotherapy has become the standard of care for breast cancer patients with large tumors in order to render them operable for mastectomy or, in some cases, for lumpectomy and radiation therapy. Building on this theme, several large hormonal therapies are extensively investigated in the neoadjuvant setting, together with biologic correlates for response and resistance. As a further extension, neoadjuvant therapies with biologic agents are now too, being investigated for biologic evidence of efficacy before large-scale clinical trials of thousands of patients are embarked on. The neoadjuvant setting is especially attractive for these studies for several reasons including early assessment of response to therapy, biopsiable access to the primary tumor, and considerable reduced sample sizes compared to those required in the adjuvant setting. In addition, clinical response to neoadjuvant chemotherapy is a validated surrogate marker for improved survival. It may be used to test the overall efficacy of neoadjuvant treatment regimens and mirrors the effect of therapy on micrometastases setting. In a recent study, good clinical response to neoadjuvant chemotherapy was the only independent variable, by multivariate analysis, associated with decreased risk of death.

GW572016 is a new and promising dual tyrosine kinase inhibitor against HER1/2. Hundreds of patients were treated in phase I and II studies world-wide and results indicate that this reversible, oral small molecule is generally well-tolerated. Studies of neoadjuvant Trastuzumab indicate that HER2 interference leads to significant tumor regression even after 3 weeks of monotherapy. We aim to extend these findings with a novel agent, GW572016 that may be more effective, especially from its in vitro data, and to discover the true response rate to inhibiting HER1/2 signal transduction in breast cancer patients.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be female.
2. Signed informed consent.
3. Only subjects with Stage IIIa, IIIb, IIIc, or IV disease should be enrolled in this trial. Locally advanced breast cancers of clinical and or radiologic size greater than or equal to 3 cm, or primary breast cancers with concomitant gross metastatic disease.
4. HER2 overexpressing tumors defined as HercepTest score of 3+, or > 10% cells moderately or strongly HER2 positive by other methods, or semi-quantitative score of >5 (in Dr. Allred's laboratory) or gene amplified.
5. Negative serum pregnancy test (beta-HCG) within 7 days of starting study, if of child-bearing potential.
6. Kidney and liver function tests - all within 1.5 times the institution's upper limit of normal.
7. Performance status (WHO scale) <2 and life expectancy >6 months.
8. Age >18 years.
9. No brain or leptomeningeal disease.
10. No previous or current malignancies at other sites within the last 5 years, with exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.

Exclusion Criteria:

1. Pregnancy or unwillingness to use a reliable contraceptive method in women of child-bearing potential.
2. Severe underlying chronic illness or disease.
3. Cardiomyopathy or baseline LVEF <50%.
4. Other investigational drugs while on study.
5. Severe or uncontrolled hypertension, history of congestive heart failure or severe coronary arterial disease.
6. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The primary end point of this study is clinical efficacy of GW572016 in treatment naïve patients with locally advanced breast cancer. | 3 years

SECONDARY OUTCOMES:
The secondary end points would be the biologic correlative of relevant biomarkers. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Royce, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- UNM CRTC, Albuquerque, New Mexico, United States